CLINICAL TRIAL: NCT02202408
Title: A Phase I, Double-blind, Randomized, Placebo-controlled, Single-Dose Escalation, First-in-human Clinical Trial to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SKI2670
Brief Title: Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of SKI2670
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SKI2670_EMSD_I_2013
Record Dates: First submitted 2014-07-16; First posted 2014-07-29 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2016-08

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — TU2670

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SKI2670 (Experimental): Single-dose escalation/ Subjects received an oral single dose of SKI2670 capsule by dosing group
  -Dosing Group 1, Dosing Group 2, Dosing Group 3, Dosing Group 4
  Interventions: Drug: SKI2670
- Placebo (Placebo Comparator): Subjects received an oral single dose of placebo capsule matched to the SKI2670 dose (Placebo for SKI2670)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SKI2670 — Oral, Single Dose
  Other Names: N/A(only SKI2670)
  Arms: SKI2670
Drug: Placebo — Same shape as the experimental drug
  Other Names: N/A(only 1 Placebo)
  Arms: Placebo

SUMMARY:
In this Phase I study, the primary objective is to investigate the safety and tolerability of SKI2670 after oral administration in healthy female subjects. And secondary objective is to investigate the pharmacokinetics and pharmacodynamics of SKI2670 after oral administration in healthy female subjects.

DETAILED DESCRIPTION:
In this Phase I study, the primary objective is to investigate the safety and tolerability of SKI2670 after oral administration in healthy female subjects.

Secondary objective is to investigate the pharmacokinetics and pharmacodynamics of SKI2670 after oral administration in healthy female subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 20 years of age and older
2. Weight between 40kg~70kg
3. Women who agreed using double contraception method and spermicide, avoiding breast-feeding for at least 30days after IP(investigational product) dosing
4. A history of regular menstrual cycles (cycle: 28±7day, duration: 2~7day) for at least 2 years and a positive ovulation test between day 11 and 21 in the preceding menstrual cycle of IP(investigational product) dosing

Exclusion Criteria:

1. Women who are pregnant or serum/urine hCG(human chorionic gonadotropin) positive or breast-feeding
2. A history of breast cancer, genital cancer or any estrogen dependent tumor
3. Specified or unspecified diagnosed infertility or history of natural abortion over three times
4. A history of taking other Investigational product within 60days before screening visit or taking ETC drug(Ethical drugs), oriental medicine or OTC drugs(Over-the-Counter drugs) within 14days before screening visit
5. Clinically significant Gynecological disease identified by ultrasonography including estrogen dependent tumor or lesion, sever inflammation or synechia
6. AST(Aspartate aminotransferase), ALT(Alanine aminotransferase) ≥ 2.5 times the upper limit of normal
7. QTc > 450ms on electrocardiogram result

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From day 1 to day 16~26D after a single oral dose.
  All participants who ever were administered with investigational product are assessed.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of SKI2670 | 0h(pre-dose), 10min, 20min, 30min, 45min, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h
  Peak Plasma Concentration (Cmax) of SKI2670
Area Under Curve (AUC) of SKI2670 | 0h(pre-dose), 10min, 20min, 30min, 45min, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h
  Area Under Curve (AUC) of SKI2670
Concentration Change from Baseline(%) of Luteinizing Hormone (LH) | day -1, 0h(pre-dose), 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 30h, 36h, 48h, 72h, day 7~12D, 16~26D
  Concentration Change from Baseline(%) of Luteinizing Hormone (LH)

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, MD,PhD, Study Chair — Asan Medical Center Department of Clinical Pharmacology and Therapeutics
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Han S, Cho YS, Yoon SK, Lim KS, Cho SH, Kim J, Choe S, Jung J, Ghim JL, Choi S, Lee M, Kim SM, Kim HT, Lim HS, Yoon Shim J, Bae KS. First-in-Human, Double-Blind, Randomized Controlled Trial of an Oral Dose of GnRH Antagonist TU2670 in Healthy Women. J Clin Endocrinol Metab. 2021 Mar 8;106(3):e1111-e1120. doi: 10.1210/clinem/dgaa939. PMID 33347565